CLINICAL TRIAL: NCT05090618
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: The Role of Genetic Factors in the Development of Myocardial Infarction in the Kazakh Population
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Head of the Laboratory of Experimental Medicine, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1187
Record Dates: First submitted 2021-09-25; First posted 2021-10-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Heart Attack
Keywords: GWAS
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: Patients with Heart Attack
  Interventions: Genetic: DNA analysis
- Control group: Patients without Heart Attack
  Interventions: Genetic: DNA analysis

INTERVENTIONS:
Genetic: DNA analysis — GWAS

SUMMARY:
This is a GWAS study that aims to identify possible candidate genes associate to heart attack by exploring single nucleotide polymorphism (SNP) in a group of heart attack, in the Kazakh population. The investigators hypothesize that the careful phenotyping of the subject sand matching with increase the power to find SNP significantly associate with heart attack

DETAILED DESCRIPTION:
A genome-wide association study (GWAS) is an approach used in genetics research to associate specific genetic variations with particular diseases. The method involves scanning the genomes from many different people and looking for genetic markers that can be used to predict the presence of a disease. Once such genetic markers are identified, they can be used to understand how genes contribute to the disease and develop better prevention and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Persons of Kazakh nationality
* Age up to 59 years inclusive at the time of primary myocardial infarction
* Myocardial infarction was established in accordance with the EOC criteria: An increase and / or decrease in the level of cardiac troponin must be combined with at least one of the following: • Symptoms of myocardial ischemia • Newly occurring ischemic changes on the ECG • The appearance of a pathological Q wave • Identification according to imaging data methods of new areas of non-viable myocardium, or new areas of local contractility disorders of presumably ischemic etiology • Detection of a thrombus in the coronary arteries according to coronary angiography
* Presence of coronary angiography
* Persons able and willing to provide written informed consent;

Exclusion Criteria:

* Age at primary myocardial infarction 60 years and older
* Heart defects, congenital and acquired
* Non-ischemic cardiomyopathies
* Autoimmune diseases
* Diabetes mellitus at the time of development of primary myocardial infarction
* Terminal stages of renal and hepatic failure

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: KAZAKH POPULATION
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
number of SNPs associated with Heart Attack | 1 year
  Using GWAS to identify candidate genes associate with Heart Attack

CONTACTS AND LOCATIONS:
Overall Officials: Aisulu Mussagaliyeva, PhD, Study Director — Research Institute of Cardiology and Internal Medicine; Roza Kuanyshbekova, Study Director — Research Institute of Cardiology and Internal Medicine
Locations (1):
- Kazakhstan, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided